CLINICAL TRIAL: NCT00938457
Title: A Phase I/II Dose-Finding Study of Single-Fraction Stereotactic Body Radiotherapy (SF-SBRT) for the Treatment of Liver Metastases
Brief Title: Stereotactic Radiation Therapy in Treating Patients With Liver Metastases
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0941; MC0941 (Other: Mayo Clinic Cancer Center); 09-000020 (Other: Mayo Clinic IRB); NCI-2009-01150 (Registry Identifier: NCI's CTRO)
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Results first posted 2012-07-09 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2015-10

CONDITIONS: Unspecified Adult Solid Tumor
Keywords: protocol specific
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients undergo either percutaneous placement of metallic fiducial markers within the liver or respiratory-correlated cone-beam computed tomography for stereotactic targeting and planning. Patients then undergo single-fraction stereotactic body radiotherapy over approximately 1 hour within 1 week of the marker placement.
  Interventions: Radiation: stereotactic radiation therapy; Procedure: implanted fiducial-based imaging; Procedure: cone-beam computed tomography

INTERVENTIONS:
Radiation: stereotactic radiation therapy — Patients undergo stereotactic body radiation therapy
Procedure: implanted fiducial-based imaging — radiation therapy treatment planning
Procedure: cone-beam computed tomography — radiation therapy treatment planning

SUMMARY:
RATIONALE: Stereotactic radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

PURPOSE: This phase I/II trial is studying the side effects and best dose of stereotactic radiation therapy in treating patients with liver metastases.

DETAILED DESCRIPTION:
OUTLINE: This is a phase I/II, dose-escalation study.

Phase I: Patients undergo either percutaneous placement of metallic fiducial markers within the liver or respiratory-correlated cone-beam computed tomography for stereotactic targeting and planning. Patients then undergo single-fraction stereotactic body radiotherapy over approximately 1 hour within 1 week of the marker placement.

Phase II: Patients undergo treatment as in phase I at the maximum tolerated dose. After completion of study treatment, patients will be followed at weeks 4 and 12 and then every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation (any histology except lymphoma, leukemia, or hepatocellular carcinoma) of at least one liver lesion that is synchronous to the primary diagnosis of malignancy or metachronous as a recurrence/metastasis or as a failure following previous therapy (except radiotherapy).
* One to three metastatic liver lesions =< 5 cm in dimension.
* Intrahepatic cholangiocarcinoma is acceptable for inclusion.
* Zubrod Performance Status (PS) 0 or 1.
* Please contact study investigator and/or consult protocol document for specific details on laboratory criteria.
* Life expectancy >= 12 weeks.
* MELD (Model for End-Stage Liver Disease) score =< 16.
* >= 1000 cc of uninvolved liver parenchyma as determined by the treating physician.
* Determination that the patient is medically inoperable and/or unwilling to undergo liver resection in patients with colorectal carcinoma histology.
* Provide informed written consent.
* Willingness to return to Mayo Clinic Rochester for follow-up.

Exclusion Criteria:

* Pregnant women.
* Nursing women.
* Men or women of childbearing potential or their partners who are unwilling to employ adequate contraception.
* Co-morbid systemic illnesses or other severe concurrent disease, defined as those which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be HIV positive.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm =< 7 days prior to registration.
* Administration of chemotherapy within 2 wks prior to or 2 wks following SF-SBRT.
* Prior radiation therapy to the liver Untreated malignant biliary obstruction (patients treated successfully with stenting are eligible).
* Current diagnosis of hepatocellular carcinoma

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-07; Primary Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Miller, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three patients were recruited at Mayo Clinic between January 2010 and May 2010.
Pre-assignment Details: This was a phase I/II trial. A total of 3 participants were accrued, all to the phase I portion. This trial was terminated due to poor accrual. No patients were accrued to the phase II portion. No results from the phase II portion are available.
Period: Overall Study
Arm/Group | Arm I
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 60 [43 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Determination of the Maximum Tolerated Dose (MTD) of Single-fraction Stereotactic Body Radiation Therapy (SF-SBRT) in Hepatic Metastases.
Time Frame: 2 months
Population: Not enough patients were accrued to the Phase I portion to determine the MTD.
Arm/Group | Arm I
Number analyzed (Participants) | 0

2. Primary Outcome: Determine the Minimum Effective Dose (MED) Necessary for Durable Local Control, Defined as the Dose Level at Which Local Control (LC) is >= 80% at 1 Year. (Phase II)
Description: LC is defined as no evidence of disease progression within the volume treated to prescription dose (i.e. PTV) for a specific lesion. The development of new intrahepatic metastases sites outside of the PTV will not be considered local failures.
Time Frame: At 1 year
Population: No patients were accrued to the Phase II portion.
Arm/Group | Arm I
Number analyzed (Participants) | 0

3. Secondary Outcome: Toxicity and Adverse Events Profile (Phase I)
Description: Number of patients with a grade >= 3 adverse event.
  Adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.
  Description of Grades:
  Grade 1: Mild Grade 2: Moderate Grade 3: Severe Grade 4: Life-threatening Grade 5: Death
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 3
participants | 0

4. Secondary Outcome: Patient Clinical Response and Treatment Effects on Blood Chemistry and Hepatic Function Markers (Phase I)
Time Frame: Up to 2 years
Arm/Group | Arm I
Number analyzed (Participants) | 0

5. Secondary Outcome: Radiographic Response Rate (Phase II)
Time Frame: Up to 2 years
Population: No patients were accrued to the Phase II portion.
Arm/Group | Arm I
Number analyzed (Participants) | 0

6. Secondary Outcome: Local Control (LC) Cumulative Incidence Rates (Phase II)
Time Frame: 3 and 6 months and 1, 2, and 5 years
Population: No patients were accrued to the Phase II portion.
Arm/Group | Arm I
Number analyzed (Participants) | 0

7. Secondary Outcome: Median Time to Progression of Treated Tumors (Phase II)
Time Frame: Up to 5 years
Population: No patients were accrued to the Phase II portion.
Arm/Group | Arm I
Number analyzed (Participants) | 0

8. Secondary Outcome: Refinement of Toxicity and Adverse Events Profile (Phase II)
Time Frame: Up to 2 years
Population: No patients were accrued to the Phase II portion.
Arm/Group | Arm I
Number analyzed (Participants) | 0

9. Secondary Outcome: Refinement of Patient Clinical Response and Treatment Effects on Blood Chemistry and Hepatic Function Markers (Phase II)
Time Frame: Up to 2 years
Population: No patients were accrued to the Phase II portion.
Arm/Group | Arm I
Number analyzed (Participants) | 0

10. Secondary Outcome: Evaluation of Cause of Death (Phase II)
Time Frame: Up to 5 years
Population: No patients were accrued to the Phase II portion.
Arm/Group | Arm I
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=3)
Pericarditis (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Bilirubin (Investigations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes